CLINICAL TRIAL: NCT02071563
Title: Food Aid Quality Review Phase II Effectiveness Study: Preventing MAM and Stunting in Burkina Faso
Brief Title: Effectiveness and Cost-Effectiveness of Four Formulations of Food Supplements for the Prevention of Wasting and Stunting in Burkina Faso
Acronym: FAQR-Burkina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); ACDI/VOCA (Other); Save the Children (Other); Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AID-016-Burkina Faso
Record Dates: First submitted 2013-09-23; First posted 2014-02-26 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Child Malnutrition
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CSB14 (Active Comparator): Isocaloric amount and cost-effectiveness of CSB14 (with whey protein concentrate and enhanced micronutrient profile), prepared with fortified vegetable oil (FVO).
  Interventions: Dietary Supplement: CSB14
- RUSF1 (Active Comparator): Isocaloric amount and cost-effectiveness of Ready-to Use Supplementary Food 1(RUSF1), USAID's Lipid-Based Nutrient Supplement (LNS) product
  Interventions: Dietary Supplement: RUSF1
- SC+ (Active Comparator): Isocaloric amount and cost-effectiveness of Supercereal Plus (SC+), the FBF used by WFP, which has an enhanced nutrient profile, dairy ingredient (non-fat dry milk), and oil already embedded into the flour
  Interventions: Dietary Supplement: SC+
- CSB+ (No Intervention): Isocaloric amount and cost-effectiveness of Supercereal/CSB+ prepared with FVO.

INTERVENTIONS:
Dietary Supplement: CSB14
  Arms: CSB14
Dietary Supplement: RUSF1
  Arms: RUSF1
Dietary Supplement: SC+
  Arms: SC+

SUMMARY:
This research will serve as a follow-up on the review of Title II commodities performed by the Food Aid Quality Review at Tufts University in October 2011. The study in Burkina Faso will test the relative effectiveness and cost effectiveness of four supplementary foods in the prevention of MAM and stunting in normal programmatic settings.

The aims of this study are to:

1. To compare the effectiveness of four alternative supplementary food commodities in preventing stunting and wasting, and promoting linear growth in children 6 - 23 months in the context of a preventive supplementary feeding program in Burkina Faso.
2. To estimate the relative cost of implementing the supplementary feeding program using each commodity
3. To estimate the relative cost/effectiveness of implementing the program using each commodity.

DETAILED DESCRIPTION:
Phase II of FAQR in Burkina Faso will assess the recommended improvements in the four arms of the study: CSB14 prepared with FVO, RUSF1, CSB+, and SC+.

The study will be a cluster-randomized, effectiveness trial. The study will use a mixed method technique of quantitative and qualitative data collection. The design of the study is quasi-experimental: food distribution sites (FDPs) (and the communities they serve) will be grouped into four clusters that are geographically contiguous with each other and sufficiently distant from each other so that the Beneficiaries are unlikely to have contact with each other. The four groups of food distribution points will be randomly assigned to one of four arms, defined by the specific food to be provided:

1. Corn Soy Blend 14 (CSB14) (with whey protein concentrate and enhanced micronutrient profile), prepared with fortified vegetable oil (FVO); 75g CSB14/day, 22.5g FVO/day
2. Ready-to use supplementary food 1 (RUSF1); 100g RUSF/day
3. Super Cereal Plus (SC+)( has an enhanced nutrient profile, non-fat dry milk, and oil already embedded into the CSB); 122g SC+/day
4. Corn Soy Blend Plus (CSB+) prepared with FVO; 75g CSB+/day, 22.5g FVO/day The CSB+ arm will act as a control

The intervention is implemented using the food distribution points providing supplementary food (CSB14, CSB+, RUSF, SC+) to children once they reach six months of age, and children from 6 to 23 months. This study will enroll all children as they turn six months of age and follow them through their 23rd month of age. Variables to be tracked include: age, sex, arm of study/commodity received ,Mid-Upper Arm Circumference (MUAC), height for age, weight for age, weight for height, month-to-month linear growth and weight gain, incidence of stunting (height for age below -2 Standard Deviations (SD)), incidence of wasting (weight for height below - 2 SD).

At 24 months, children stop receiving supplementary food. The study will continue to monitor these variables for at least an additional 6 months (through the age of 30 months).

The study will collect information on the following additional variables from Beneficiary Mothers/Caretakers, Health and Nutrition Promoters (HNPs), Community Health Agents (CHAs), store owners who sell products comparable to those distributed, and PVO staff members.

* Mothers' knowledge, attitude, and practices with respect to compliance with instructions about the preparation and use of the supplementary food
* Time and money costs to Beneficiary Mothers/Caretakers of participating in the feeding program
* Household Characteristics
* Environmental characteristics
* Community characteristics
* Perceived barriers and factors facilitating Title II program effectiveness
* Logistics and cost of procuring, warehousing and distributing the food to the food distribution point

Data Collection Time Points Data collection will be ongoing. It is expected that in order to reach our sample size, the study will need to enroll children on a rolling basis when they turn 6 months old for one year. All children will receive a food ration for 18 months, until they turn 2 years old. During this time period, the study will collect growth measurements (height, weight, MUAC) on every enrolled child at monthly intervals.

Throughout the study, qualitative and quantitative data will also be collected from Beneficiary Mothers/Caretakers, Health and Nutrition Promoters (HNPs), Community Health Agents (CHAs), and PVO staff members as described above. We will conduct qualitative open ended interviews with PVO staff members in their professional capacities, to learn of any challenges or strengths in implementing the procurement and distribution of new commodities.

We will also randomly select a small subsample of Beneficiary Mothers/Caretakers for in-home observations. The purpose of these observations is to observe aspects of the family's preparation and consumption of the ration that they would be unlikely to be able to report during focus groups or individual interviews, because respondents may not be conscious of their actions. Examples include: giving tastes of the ration to children while it is being cooked; how quickly the ration is covered after feeding; whether children are able to take tastes of leftover rations. We would follow a commonly used model of asking families to have a guest observer stay with them for up to a week during waking hours. The observer would collect information on these aspects of preparation and consumption methods and on other observable behavior (e.g. how many times a day the ration is made, whether covered while cooking, after cooking, after serving).

We will collect a small (2 tablespoon) sample of prepared ration from all individually interviewed Beneficiary Mothers/Caretakers. This will be used for laboratory assessment of the proportion of FVO in the porridge to validate our estimates of the CSB : Oil ratio as reported by the mother.

The objective of this study is to highlight which food product best prevents stunting and MAM, in the most cost effective way, thereby ultimately affecting future effective and efficient policy in food aid programs.

ELIGIBILITY:
The subjects are as follows:

Beneficiary Children that are weighed and measured Beneficiary Mothers/Caretakers that participate in interviews, focus group discussions, and in-home observations Health and Nutrition Promoters (HNP) that participate in individual interviews and FGD Community Health Agents that participate in individual interviews PVO staff members that participate in individual interviews Village Elders/Headmen Store owners/Market Vendors that participate in individual interviews

Beneficiary Children (Children 6 -23 months old)

* Inclusion Criteria

  • Child enrolled in the ViM program to receive ration from a Food Distribution Point
* Exclusion Criteria

  * Children who are over 6 months of age when the study begins
  * Children receiving food rations from another organization (e.g. World Food Programme or UNICEF)

Beneficiary Mothers/Caretakers (Mothers/Caretakers of Children 6 -23 months old)

* Inclusion Criteria

  * Beneficiary Mother/Caretaker whose child turns 6 months old and is enrolled in ViM program to receive ration during the study period
  * Beneficiary Mother/Caretaker has no age restrictions for inclusion (Note: Mothers/caretakers will be asked to participate regardless of age and consented appropriately; it is possible some mothers may be minors)
  * Subject who is voluntarily willing to participate and indicates by signing (or marking with a thumbprint) the consent form.
* Exclusion Criteria • Beneficiary Mothers/Caretakers who participate in an interview, observation or FGD once for this study will not be eligible again for participation

Health and Nutrition Promoters (HNP) Inclusion Criteria

* HNP who covers the catchment area of the FDPs
* Subject who is voluntarily willing to participate by signing the consent form

Community Health Agents (CHA) Inclusion Criteria

* Community Health Agents serving within the catchment area for the FDPs
* Community Health Agents that have been present during the study period
* Subject who is voluntarily willing to participate and indicates by signing the consent form

PVO Staff Members Inclusion Criteria

* All staff members from ACDI/VOCA and Save the Children who are directly involved in the ViM program
* Subject who is voluntarily willing to participate and indicates by signing the consent form Exclusion Criteria
* PVO Staff members who joined too recently to have experience of the program change (new commodities)

Village Elders/Headmen Inclusion Criteria

* Village elder/headmen in study commune
* Subject who is voluntarily willing to participate and indicates by signing the consent form Exclusion Criteria
* Village elder/headmen whose community is not involved in the feeding program

Store Owners/Market Vendor Inclusion Criteria

* Store owner/market vendor in study communes who trades in the relevant products (food vendors)
* Subject who is voluntarily willing to participate and indicates by signing the consent form Exclusion Criteria
* Vendors who do not sell food.

The withdrawal/termination criterion for this study is not applicable as the subject's participation will not be terminated by the investigator, and there are no necessary precautions applied to those who withdraw.

Study subjects may not participate in another research study that provides supplementary food as a food ration to children between 6-23 months.

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6039 (Actual)
Dates: Start 2014-03; Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Incidence of MAM and Stunting | Monthly for 18 months
  Primary outcomes to be measured are incidence of MAM and incidence of stunting during the 18 months of preventive supplementation (age 6 months to 23 months).
  Stunting will be defined as less than -2 SD of Height-for-Age Z-score and MAM will be defined as less than -2 SD Weight-for-Height (length) Z-score

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice L Rogers, PhD, Principal Investigator — Tufts University
Locations (1):
- Kaya, Sanmatenga, Burkina Faso

REFERENCES:
- [Derived] Cliffer IR, Naumova EN, Masters WA, Perumal N, Garanet F, Rogers BL. Peak timing of slowest growth velocity among young children coincides with highest ambient temperatures in Burkina Faso: a longitudinal study. Am J Clin Nutr. 2024 Feb;119(2):393-405. doi: 10.1016/j.ajcnut.2023.09.021. Epub 2023 Dec 29. PMID 38309828
- [Derived] Cliffer IR, Masters WA, Perumal N, Naumova EN, Zeba AN, Garanet F, Rogers BL. Monthly measurement of child lengths between 6 and 27 months of age in Burkina Faso reveals both chronic and episodic growth faltering. Am J Clin Nutr. 2022 Jan 11;115(1):94-104. doi: 10.1093/ajcn/nqab309. PMID 34637506
- [Derived] Shen Y, Cliffer IR, Suri DJ, Langlois BK, Vosti SA, Webb P, Rogers BL. Impact of stakeholder perspectives on cost-effectiveness estimates of four specialized nutritious foods for preventing stunting and wasting in children 6-23 months in Burkina Faso. Nutr J. 2020 Feb 27;19(1):20. doi: 10.1186/s12937-020-00535-x. PMID 32106840
- [Derived] Cliffer IR, Nikiema L, Langlois BK, Zeba AN, Shen Y, Lanou HB, Suri DJ, Garanet F, Chui K, Vosti S, Walton S, Rosenberg I, Webb P, Rogers BL. Cost-Effectiveness of 4 Specialized Nutritious Foods in the Prevention of Stunting and Wasting in Children Aged 6-23 Months in Burkina Faso: A Geographically Randomized Trial. Curr Dev Nutr. 2020 Jan 23;4(2):nzaa006. doi: 10.1093/cdn/nzaa006. eCollection 2020 Feb. PMID 32072130
- [Derived] Langlois BK, Cliffer IR, Nikiema L, Suri DJ, Garanet F, Shen Y, Zeba AN, Walton SM, Lanou HB, Webb P, Rogers BL. Factors that May Influence the Effectiveness of 4 Specialized Nutritious Foods in the Prevention of Stunting and Wasting in Children Aged 6-23 Months in Burkina Faso. Curr Dev Nutr. 2020 Jan 6;4(2):nzaa002. doi: 10.1093/cdn/nzaa002. eCollection 2020 Feb. PMID 31998858